CLINICAL TRIAL: NCT01250132
Title: Are Ante-hypophyseal Dysfunctions in the Acute Phase of Moderate to Severe Traumatic Brain Injury Predictive of Long-term Ante-hypophyseal Sequelae in Children?
Brief Title: Ante-hypophyseal Dysfunctions in Children Following Moderate to Severe Traumatic Brain Injuries
Acronym: Endoc-TC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2010.599
Record Dates: First submitted 2010-11-25; First posted 2010-11-30 (Estimated); Last update posted 2019-09-04 (Actual); Status verified 2019-08

CONDITIONS: Moderate to Severe Traumatic Brain Injury
Keywords: Traumatic brain injury; Paediatrics; Hypopituitarism
MeSH Terms: conditions — Brain Injuries, Traumatic; Hypopituitarism | interventions — Biological Products

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Moderate to severe Traumatic Brain Injury (Other): Assessment of hypopituitarism. Blood tests at different moments:
  * day 0
  * when leaving intensive care unit
  * month 3
  * month 12
  Interventions: Other: Biological and behavioral explorations

INTERVENTIONS:
Other: Biological and behavioral explorations — Blood dosages:
  * biochemistry
  * pituitary gland
  * somatotropic axis
  * corticotropic axis
  * gonadotropic axis
  * thyrotropic axis
  * antidiuretic axis
  Questionnaires and scales (quality of life, Vineland Adaptive Behavior Scales (VABS)-II)

SUMMARY:
Annual incidence of severe traumatic brain injuries (TBI) varies from 180 to 300 out of 100.000. Mortality or severe sequelae risk is increased 8 fold after a TBI. Studies in adults showed an ante-hypophyseal deficit in 28 to 68 % of patients with a TBI. The most common deficit is Growth Hormone Deficit (GHD); followed by gonadotropic and corticotropic (AdrenoCorticoTropic Hormone (ACTH)) insufficiencies. Thyrotropic deficits (Thyroid-Stimulating Hormone (TSH)) are less frequent. From a pathophysiological point of view, the lesional mechanism responsible for hypopituitarisms would be a damage of hypophyseal vessels or hypothalamic-pituitary vessels. The frequency of pituitary deficits and the potential beneficial effects of replacement therapy on quality of life, tiredness, loss of energy and productivity, justify the systematic detection of the deficits in patients with moderate to severe TBI.

Study hypotheses :

At the present time, the lack of data in children does not give us the opportunity to affirm that one part of the symptoms showed by children with post-TBI neuropsychological sequelae, are linked to pituitary deficiency and that they can be improved with a replacement therapy.

Firstly, it is essential to better understand the natural history of post-TBI pituitary deficiencies, studying the connexion between observed deficiencies in acute and late phase of sequelae.

ELIGIBILITY:
Inclusion Criteria:

* children from 2 months to 16 years
* in the intensive care unit
* TBI : moderate (Glasgow Coma Scale (GCS) between 9 and 12) to severe (GCS <9), whatever the mechanism involved
* informed consent form signed by parents

Exclusion Criteria:

* obesity (Body Mass Index (BMI) > 97th percentile for the age)
* patient already under replacement therapy.
* patient taking AntiEpileptic Drugs (AEDs)
* patient with long-term systemic corticotherapy
* history of neurological disease or learning difficulties
* no covered by a national health insurance

Ages: 2 Months to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 110 (Actual)
Dates: Start 2010-10 (Actual); Primary Completion 2018-04-13 (Actual); Study Completion 2018-04-13 (Actual)

PRIMARY OUTCOMES:
Study the link between pituitary deficiencies highlighted at the acute phase and one year after moderate to severe TBI. | 12 months after inclusion

SECONDARY OUTCOMES:
Study the association between pituitary deficiencies highlighted at the acute phase, 3 months and 1 year after moderate to severe TBI, globally and per deficiency category. | day0, when leaving intensive care unit, month3 and month12
Identify the other risk factors of deficiency, during the acute phase and the tardive phase i.e. signs of gravity of the TBI, type of cerebral lesion, age, lesional mechanism. | day0, when leaving intensive care unit, month3 and month12
Study the correlation between corticotropic deficiencies and post-hypophysis insufficiencies during the acute phase and the hemodynamic instability over the first 3 days after the TBI | day0 to day3
Compare the level and the type of behavioural and neuropsychological sequelae in children suffering from a TBI, with and without hypopituitarism. | day0, when leaving intensive care unit, month3 and month12

CONTACTS AND LOCATIONS:
Overall Officials: Etienne JAVOUHEY, MD, PhD, Principal Investigator — Hospices Civils de Lyon
Locations (2):
- France (2):
  - CHU de Grenoble, Grenoble
  - Hospices Civils de Lyon, Lyon